CLINICAL TRIAL: NCT05349929
Title: Comparison of the Analgesic Effect of Bromelain and Ibuprofen on Pain After Root Canal Treatment(A Clinical Trial Study)
Brief Title: Analgesic Effect of Anahil and Ibuprofen on Pain After Root Canal Therapy in Patients With Pulpitis of the Molars in Qazvin(a City in Iran)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mona Esfahani, Dentistry Student, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1111
Record Dates: First submitted 2022-04-05; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Irreversible Pulpitis
MeSH Terms: interventions — Root Canal Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ibuprofen (Experimental): Ibuprofen(Gelofen) 400mg capsules, Dana pharma company, every 6hours
  Interventions: Drug: Gelofen (generic name of Ibuprofen in Iran); Procedure: Root Canal Therapy
- Anahil (Experimental): Bromelain(Anahil) 200 mg capsules, Permon Amin Health Company,every 6hours
  Interventions: Drug: Anahil ( generic name of Bromelain in Iran); Procedure: Root Canal Therapy

INTERVENTIONS:
Drug: Gelofen (generic name of Ibuprofen in Iran) — Gelofen capsules, 400mg Ibuprofen, Dana pharma company, every 6hours
  Arms: Ibuprofen
Drug: Anahil ( generic name of Bromelain in Iran) — Anahil capsules,200 mg Bromelain, Permon Amin Health Company,every 6hours
  Arms: Anahil
Procedure: Root Canal Therapy — all the participants go under RCT.

SUMMARY:
Hypothesis:

0: The analgesic effect of Ibuprofen and Anahil would be the same in reducing the pain after root canal therapy.

1: Ibuprofen shows higher potency to reduce the pain after root canal therapy.

1: Anahil shows higher potency to reduce the pain after root canal therapy.

1. combination of the Anahil and Ibuprofen would have more effective results in reducing the pain post endodontic treatment.

DETAILED DESCRIPTION:
Patients will be selected from those who are referred to receive root canal therapy for the mandibular first molars with irreversible pulpitis.

The current research and all the procedures will be done in a private dental clinic in Qazvin, Iran by a single endodontist.

72 Patients who will meet our study demands and criteria would be qualified to enter the study and will sign the informed consent form explaining the study circumstances and its possible risks.

Patient information sheet includes dental, medical and drug history and demographic information will be obtained as well. Radiographic examination includes the amount of caries, root curvature, periapical and hard tissue situation, dental pulp vitality tests including Electrical Pulp Test(EPT) and thermal tests (heat and cold) and periapical tests consisting of percussion and palpation would be recorded. The patients would be divided randomly in Ibuprofen and Anahil groups, these drugs would be put in the same shape and appearance by a pharmacist and named as A and B respectively. Anahil capsules containing 200 mg of bromelain, Permon-Amin Health Company, Gelofen 400mg capsules, Dana-Pharma company:The pre procedure pain of the patients would be asked and recorded by Visual Analogue Scale(VAS), a 100 mm long ruler which has no numeration by means of enhancing the accuracy and minimizing the failure. Standard Infra alveolar nerve(IAN) direct block will be done by injection of 1.8ml of lidocaine 2% containing 1:100000 epinephrine with a long 32mm gauge 27 needle. The efficiency of Inferior Alveolar Nerve block injection will be examined with the numbness of inferior lip. Supplementary anesthesia (like intrapulpal or Periodontal Ligament(PDL) anesthesia) will be used if the pain is still remained after 15 minutes. After tooth isolation with rubberdam, caries removal, access cavity and tooth preparation will be done. Length determination will be performed with the help of periapical radiography and apex locator. Cleaning and shaping will be done. Normal Saline and hypochlorite 2% will be used as intracanal irrigants. The canals will then be dried and gutted laterally with gutta-percha and AH+ sealer. A cotton pellet will be placed in the access cavity. Temporary restoration will be applied after occlusal reduction and the occlusion will be checked. No intracanal medicament will be placed. In this triple blinded study, patients will be given A and B drugs (36 patients in each group, equal in gender) with medications order randomly and will be followed 6, 12, 24 and 48 hours after endodontics treatment to report the pain score with VAS and the number of supplementary dosage of Ibuprofen with the time that they have consumed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients report spontaneous pain of the first molar of mandible ranging from 50 to 100 mm on a VAS (0-100 mm)
2. The dental pulp's condition is irreversible pulpitis and the tooth is reparable and need the root canal therapy
3. No evidences of any lesions and lucency, PDL widening, loss of lamina dura in radiographic examination
4. Patients aged 20 to 50 years from both genders
5. Patients are not pregnant or breast-feeding
6. Healthy periodontal status (no evidences of aggressive/chronic periodontal diseases)
7. No history of any systemic diseases (specially gastrointestinal and coagulation disorders)
8. No history of allergic reaction to food nutrients (specially pineapple, celery, carrot, and fennel), NSAIDs and lidocaine
9. No history of consuming the drugs interfere with NSAIDs, lidocaine and anticoagulants
10. No use of other analgesic drugs within the last 6 hours
11. Existence of no large restorations or crowns in treated tooth
12. patients have no extreme fear of dental procedure
13. Teeth with no evidence of infection or sinus tract
14. Patients did not a previous RCT

Exclusion Criteria:

1. Patients who leave the study because of any reasons
2. Special anatomy of teeth (extra canals, severe root curvature, calcifications, open apex, C shape, fractures,..)
3. Patients who are not able to tolerate the single-session treatment (time, tooth's situation,..)
4. If the aspiration through IAN block injection is positive
5. If the diagnosis of pulp status has changed to partial necrosis during access cavity preparation

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
pain severity | 0 hour (before root canal treatment)
  Visual Analogue Scale
pain severity | 6 hours after root canal treatment
  Visual Analogue Scale
pain severity | 12 hours after root canal treatment
  Visual Analogue Scale
pain severity | 24 hours after root canal treatment
  Visual Analogue Scale
pain severity | 48 hours after root canal treatment
  Visual Analogue Scale
need of supplemental dosage of Ibuprofen | 6 hours after root canal treatment
  By asking the numbers of consuming capsules
need of supplemental dosage of Ibuprofen | 12 hours after root canal treatment
  By asking the numbers of consuming capsules
need of supplemental dosage of Ibuprofen | 24 hours after root canal treatment
  By asking the numbers of consuming capsules
need of supplemental dosage of Ibuprofen | 48 hours after root canal treatment
  By asking the numbers of consuming capsules

CONTACTS AND LOCATIONS:
Overall Officials: Mahsa Esfehani, Ms, Study Director — associate professor of oral medicine of Qazvin University Of Medical Sciences